CLINICAL TRIAL: NCT00198783
Title: Real-Time Assessment of Food Craving, Use, and Triggers During Outpatient Treatment of Obesity: A Development and Feasibility Study
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Other Study IDs: NIDA2005-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Obesity; Weight Maintenance
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study will assess the feasibility of utilizing real-time data monitoring in future clinical trials of weight control medications and other treatment modalities, along with the feasibility of distinguishing different types of relapses over 16 weeks: There will be 4 weeks of high-intensity EMA and 12 weeks of low-intensity EMA. Each participant will be in the study for 52 weeks with 20 visits, including follow-up visits.

DETAILED DESCRIPTION:
* Interested persons, recruited by advertisement and screened by telephone (Appendix B), will report to the Johns Hopkins Bloomberg School of Public Health for in-person screening. At the screening session, we will obtain informed consent, HIPAA consent, medical-history information (including current medications, alcohol, and cigarette use), and baseline measurements of bioelectrical impedance (BIA-body composition testing), blood pressure, pulse, body weight, and waist and hip circumference. Individuals will also be screened with established instruments for eating-disorder symptoms (Appendix C), and depression (Appendix D).
* After deemed eligible, subjects will be prescribed an individualized diet and exercise program at Visit 2 (Week 0). Additional questionnaires to be done at this visit: Restraint Scale, Three-Factor Eating Questionnaire (TFEQ), and Reasons for Dieting (Appendix E).
* At the same visit, each participant will be issued a PDA and trained in its use as an Electronic Diary (ED). Participants will be expected to carry their PDAs at all times.
* A 4-week period of high-frequency monitoring will begin immediately: random prompts to initiate recordings will occur 0-5 times per day for 4 weeks. Participants must respond to at least 85% of all random prompts within 15 minutes. Participants will also initiate recordings whenever they have just experienced an urge to eat, or whenever they have actually eaten.
* Participants will be randomly assigned to a Group condition or a No-Group condition.
* In the Group condition, participants will attend 10 group meetings, starting at Week 2 (Visit 4), to strengthen diet-adherence and lapse-management skills. Group meetings will be held once every week for the first 5 weeks, and once every other week for the next 11 weeks.
* In the No-group condition, participants will be given some written tips on diet adherence, but will not attend group.
* All participants must come to the clinic at scheduled times (one time per week) to upload information from the PDA to a central data source. Participants will also be weighed at these visits. This may, for some participants, coincide with the scheduled group meetings
* During Week 5-16, the frequency of EMA random prompts will be reduced to 0-2 per day.
* During Week 8 we will re-weigh the participant and reevaluate each participant's diet and exercise program to ensure a proper and safe weight-maintenance regimen. We will also record the participant's height, weight, BIA, waist and hip measurements, blood pressure, and pulse.
* A final reevaluation and weigh-in will also occur when the participant finishes the study (Week 17). We will also record the participant's height, weight, BIA, waist and hip measurements, blood pressure, and pulse
* Participants will return their PDA to the clinic at this visit.
* At Weeks 26 and 52, participants will return for a follow-up visits at which they will be re-weighed and their current diet and exercise habits will be assessed. We will also record their height, weight, BIA, waist and hip measurements, blood pressure, and pulse.
* Participants will be paid $15 each time they provide ED data for upload (up to a maximum once per week). Subjects will receive an additional $80 for completing all 16 weeks, for a possible total of $320. Additionally, participants will be paid $50 for each follow-up visit at Weeks 26 and 52. Total compensation will be $420 for completion of the entire protocol. In addition, participants will be provided compensation for paying to park at a garage at the Johns Hopkins campus.
* Participants will be removed from the study if they: behave inappropriately; lose or damage two PDAs; miss more than three scheduled clinic visits; or fail to respond within 15 minutes to more than 15% of random prompts during either phase 1 or 2 of EMA.

ELIGIBILITY:
Inclusion Criteria:

1) age between 18 and 65; 2) BMI > 30 kg/m2 prior to weight loss; 3) initial weight loss in the 12-month period prior to enrolling of at least 10% of starting body weight; 4) no more than 50% regain of that initial weight loss by the time of screening.

Exclusion Criteria:

1) Schizophrenia or any other DSM-IV psychotic disorder; history of bipolar disorder; current Major Depressive Disorder; 2) current dependence on alcohol or sedative-hypnotic, e.g. benzodiazepine (by DSM-IV criteria); 3) cognitive impairment severe enough to preclude informed consent or valid self-report; 4) medical illness that in the view of the investigators would compromise participation in research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2005-08; Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States